CLINICAL TRIAL: NCT05474573
Title: Concurrent Fluorescence and Sonographically Guided Eradication of Gliomas and Metastases Enhancing Contrast Agent in Magnetic Resonance Imaging: a Randomised, Controlled Trial
Brief Title: Concurrent Fluorescence and Sonographically Guided Eradication of Contrast-enhancing Gliomas and Metastases
Acronym: CONFLUENSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sklifosovsky Institute of Emergency Care (Other Government)
Responsible Party: Principal Investigator, Alexander Dmitriev, Neurosurgeon, MD, Sklifosovsky Institute of Emergency Care
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9c
Record Dates: First submitted 2022-07-23; First posted 2022-07-26 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Glioma, Malignant; Metastases to Brain
Keywords: contrast-enhancing glioma; brain metastasis; sonography; ultrasound; fluorescence; 5-aminolevulinic acid; 5-ALA
MeSH Terms: conditions — Glioma; Brain Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Tumor extent of resection will be assessed by radiologists blinded for the treatment arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fluorescence and Ultrasound (Experimental): Extent of tumor resection will be intraoperatively assessed using both fluorescence with 5-aminolevulinic acid and sonography
  Interventions: Device: Combined ultrasound and fluorescence-guided brain tumor resection
- Fluorescence (Active Comparator): Extent of tumor resection will be intraoperatively assessed using fluorescence with 5-aminolevulinic acid
  Interventions: Device: Fluorescence-guided brain tumor resection

INTERVENTIONS:
Device: Combined ultrasound and fluorescence-guided brain tumor resection — Surgeon intraoperatively assesses extent of tumor resection observing it's fluorescence in microscope and performing sonography
  Arms: Fluorescence and Ultrasound
Device: Fluorescence-guided brain tumor resection — Surgeon intraoperatively assesses extent of tumor resection observing it's fluorescence in microscope
  Arms: Fluorescence

SUMMARY:
Objective of the study is to determine whether combined use of intraoperative fluorescence with 5-aminolevulinic acid (5-ALA) and sonography can achieve higher rate of gross total resection of contrast-enhancing gliomas and brain metastases compared to intraoperative fluorescence with 5-ALA alone.

DETAILED DESCRIPTION:
Fluorescence-guided resection of contrast-enhancing gliomas and metastases increases extent of tumor resection. But the main drawback of this method is an inability to observe tumor fluorescence while it is covered with normal brain. Ultrasound can resolve this problem, allowing to reveal such tumor remnants. By the time there are published results of randomized control trials comparing these two technics.

Objective of the study is to determine whether combined use of intraoperative fluorescence with 5-aminolevulinic acid (5-ALA) and sonography can achieve higher rate of gross total resection of contrast-enhancing gliomas and brain metastases compared to intraoperative fluorescence with 5-ALA alone.

Participants of the study will be randomly operated using both fluorescence with 5-ALA and intraoperative ultrasound versus fluorescence with 5-ALA alone. Extent of resection will be assessed in postoperative MRI by blinded radiologists.

ELIGIBILITY:
Inclusion Criteria:

* single gliomas with contrast enhancement in preoperative magnetic resonance imaging (presumed high-grade gliomas)
* one or several brain metastases from any cancer
* newly diagnosed
* Karnofsky Performance Status 60-100%
* age 18-79 years
* performed magnetic resonance imaging with contrast enhancement

Exclusion Criteria:

* tumor spreading to corpus callosum or brainstem
* previously performed brain radiotherapy
* planned supratotal tumor resection until neurophysiologically revealed eloquent areas
* known hypersensibility to 5-aminolevulinic or to porphyrin
* hepatic or renal insufficiency
* porphyria
* pregnancy
* breast feeding

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Gross total resection (Yes or No) | within 48 hours after surgery
  No residual contrast enhancement in postoperative T1-weighted magnetic resonance imaging

SECONDARY OUTCOMES:
Extent of resection (in percents) | within 48 hours after surgery
  Extent of resection = (preoperative tumor volume - postoperative tumor volume) / preoperative tumor volume x 100
Motor function (in grades) | within 10 days after surgery
  Motor function is assessed in Medical Research Council scale
Speech function (in grades) | within 10 days after surgery
  Speech function is assessed in Hendrix scale (2017)
Karnofsky performance status (in percents) | within 10 days after surgery
  Assesses patients' possibilities to self-service in Karnofsky Performance Status scale
Cerebral complications | From admission to intensive care unit after surgery till hospital discharge, up to 365 days
  Which cerebral complications arose after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Dmitriev, MD, Principal Investigator — Sklifosovsky Institute of Emergency Care
Locations (1):
- Sklifosovsky Institute of Emergency Care, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No